CLINICAL TRIAL: NCT06562933
Title: Comparison of Efficiency of Interferential Current Application Methods in Chronic Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Serdar Kilinc, Assistant professor, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-SK-8
Record Dates: First submitted 2024-08-18; First posted 2024-08-20 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Chronic Neck Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham vacuum (Sham Comparator): Sham vacuum
  Interventions: Device: Sham vacuum
- Interferential Current Therapy Vacuum Electrodes (Active Comparator): Interferential Current Therapy Vacuum Electrodes
  Interventions: Device: Interferential Current Therapy Vacuum Electrodes
- Interferential Current Therapy Carbon-silicon Pad Electrodes (Active Comparator): Interferential Current Therapy Carbon-silicon Pad Electrodes
  Interventions: Device: Interferential Current Therapy Carbon-silicon Pad Electrodes

INTERVENTIONS:
Device: Sham vacuum — Participants will undergo a total of 10 treatment sessions over two weeks, with one session per day, five days a week. Two-channel four vacuum electrodes will be placed on the neck so that the painful area remains in the middle. The vacuum electrodes will apply continuous vacuum mode for only 10 minutes without delivering interferential current. Following the sham vacuum therapy, a hot pack will be applied to the painful neck area for 20 minutes.
  Arms: Sham vacuum
Device: Interferential Current Therapy Vacuum Electrodes — Participants will undergo a total of 10 treatment sessions over two weeks, with one session per day, five days a week. Two-channel four vacuum electrodes will be placed on the neck so that the painful area remains in the middle. Interferential current therapy with a 4000 Hz carrier frequency and 50 Hz amplitude-modulated frequency will be applied for 10 minutes using the vacuum electrodes. After the interferential current therapy, a hot pack will be applied to the painful neck area for 20 minutes.
  Arms: Interferential Current Therapy Vacuum Electrodes
Device: Interferential Current Therapy Carbon-silicon Pad Electrodes — Participants will undergo a total of 10 treatment sessions over two weeks, with one session per day, five days a week. Two-channel four carbon-silicon pad electrodes will be placed on the neck so that the painful area remains in the middle. Interferential current therapy with a 4000 Hz carrier frequency and 50 Hz amplitude-modulated frequency will be applied for 10 minutes using the carbon-silicon pad electrodes. Following the interferential current therapy, a hot pack will be applied to the painful neck area for 20 minutes.
  Arms: Interferential Current Therapy Carbon-silicon Pad Electrodes

SUMMARY:
The aim of this study is to evaluate the effects of Interferential Current Therapy on pain, disability, and quality of life in patients with chronic neck pain and to compare the effects of applying Interferential Current Therapy with vacuum electrodes versus carbon-silicon pad electrodes.

DETAILED DESCRIPTION:
Neck pain is quite common in the adult population and is a frequent reason for seeking medical attention. The prevalence of neck problems has increased with modern lifestyle changes. In individuals with neck pain, symptoms may resolve on their own within a few weeks, but approximately 30% of cases can become chronic. Neck pain lasting 1-4 weeks is considered acute; 4-12 weeks is subacute; and neck pain persisting for 12 weeks or more is considered chronic. Interferential current therapy is used in the treatment of chronic neck pain and is one of the physical therapy methods with analgesic effects. It is widely used around the world. Interferential Current Therapy can be applied using two types of electrodes: vacuum electrodes and carbon-silicon pad electrodes.The aim of this study is to evaluate the effects of Interferential Current Therapy on pain, disability, and quality of life in patients with chronic neck pain and to compare the effects of applying Interferential Current Therapy with vacuum electrodes versus carbon-silicon pad electrodes

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neck pain lasting at least 3 months
* Ages between 20 and 50 years

Exclusion Criteria:

* Patients with inflammatory or infectious diseases and those with radiculopathy or myelopathy symptoms
* Patients for whom electrotherapy is contraindicated (e.g., those with pregnancy, neurological conditions such as epilepsy, inner ear hearing aids, arrhythmias, pacemakers, active infections, skin lesions, etc.)
* Individuals with a history of malignancy, major surgery, or previous trauma
* Individuals who have received physical therapy within the last year
* Patients whose evaluation could not be completed for any reason
* Patients who do not wish to complete their evaluations for any reason

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
The Numerical Pain Rating Scale | Before treatment
  It is used to measure pain. The numerical scale for perceived pain intensity usually includes 11 numbers. The participant selects the number that best reflects their pain.In our study, participants were informed that '0' indicates no pain and '10' represents pain of unbearable intensity.
The Numerical Pain Rating Scale | 2 week after treatment
  It is used to measure pain. The numerical scale for perceived pain intensity usually includes 11 numbers. The participant selects the number that best reflects their pain.In our study, participants were informed that '0' indicates no pain and '10' represents pain of unbearable intensity.
Pressure Pain Threshold | Before treatment
  A pressure algometer (dolorimeter) is a device used for assessing pain sensitivity and measuring pressure perception.It has been proven useful in evaluating trigger points, arthritis activation, and visceral pain-pressure sensitivity. The pressure algometer consists of a metal piston with a rubber disc at the end, which has a 1 cm² surface, and is connected to a gauge that measures pressure in kilograms of force (kgf). In our study, a manual algometer (BaselineR Dolorimeter, Fabrication Enterprises, Inc, NY, USA) was used. The algometric measurement will be performed three times on the most painful point as reported by the patient and detected by palpation. The average of these three measurements will be included in the evaluation.
Pressure Pain Threshold | 2 week after treatment
  A pressure algometer (dolorimeter) is a device used for assessing pain sensitivity and measuring pressure perception.It has been proven useful in evaluating trigger points, arthritis activation, and visceral pain-pressure sensitivity. The pressure algometer consists of a metal piston with a rubber disc at the end, which has a 1 cm² surface, and is connected to a gauge that measures pressure in kilograms of force (kgf). In our study, a manual algometer (BaselineR Dolorimeter, Fabrication Enterprises, Inc, NY, USA) was used. The algometric measurement will be performed three times on the most painful point as reported by the patient and detected by palpation. The average of these three measurements will be included in the evaluation.
Neck Bournemouth Questionnaire | Before treatment
  Adapted from the Bournemouth Low Back Pain Questionnaire developed by Bolton and Humphreys in 2002, this questionnaire includes variables that must be assessed in individuals with neck pain. The content of the questionnaire covers pain intensity, the impact of pain on daily living activities and social life, anxiety and depression levels, kinesiophobia, and pain coping strategies. Each of the 7 questions is scored from 0 to 10. The highest possible score is 70, with a higher score indicating a higher level of disability.
Neck Bournemouth Questionnaire | 2 week after treatment
  Adapted from the Bournemouth Low Back Pain Questionnaire developed by Bolton and Humphreys in 2002, this questionnaire includes variables that must be assessed in individuals with neck pain. The content of the questionnaire covers pain intensity, the impact of pain on daily living activities and social life, anxiety and depression levels, kinesiophobia, and pain coping strategies. Each of the 7 questions is scored from 0 to 10. The highest possible score is 70, with a higher score indicating a higher level of disability.
Neck Disability Index | Before treatment
  The Neck Disability Index (NDI) Turkish version was used for assessing patients' disability. This index is a scale consisting of 10 questions used to evaluate how and to what extent neck pain affects the patient's daily living activities. The scale includes parameters such as pain intensity, self-care, lifting, reading, headache, concentration, driving, sleep, and social activities. Patients were asked to mark the option that best applies to them from the 6 choices provided for each parameter. Each item is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (total disability). After obtaining the total score, the value calculated according to the formula is expressed as a percentage of impairment. As the score increases, disability increases; as the score decreases, disability decreases.
Neck Disability Index | 2 week after treatment
  The Neck Disability Index (NDI) Turkish version was used for assessing patients' disability. This index is a scale consisting of 10 questions used to evaluate how and to what extent neck pain affects the patient's daily living activities. The scale includes parameters such as pain intensity, self-care, lifting, reading, headache, concentration, driving, sleep, and social activities. Patients were asked to mark the option that best applies to them from the 6 choices provided for each parameter. Each item is scored from 0 (no disability) to 5 (complete disability). The total score ranges from 0 (no disability) to 50 (total disability). After obtaining the total score, the value calculated according to the formula is expressed as a percentage of impairment. As the score increases, disability increases; as the score decreases, disability decreases.

CONTACTS AND LOCATIONS:
Locations (1):
- Abant Izzet Baysal University, Bolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No